CLINICAL TRIAL: NCT05210439
Title: Efficacy and Safety of 7 Versus 14 Days of Antibiotic Treatment for Pseudomonas Aeruginosa Bacteremia: a Multicenter, Randomized Clinical Trial (SHORTEN-2) With a DOOR / RADAR Analysis
Brief Title: Efficacy and Safety of 7 Versus 14 Days of Antibiotic Treatment for Pseudomonas Aeruginosa Bacteraemia
Acronym: SHORTEN2
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network); CIBER (Infectious diseases) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHORTEN II; 2021-003847-10 (EudraCT Number)
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bloodstream Infection
Keywords: Bacteremia; Pseudomonas aeruginosa; Bloodstream infection; DOOR / RADAR Analysis; Antimicrobial stewardship
MeSH Terms: conditions — Sepsis; Bacteremia; Pseudomonas Infections | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized 1:1 to experimental group (short-treatment arm):control group (long-treatment arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-treatment of any active antibiotic regimen (Experimental): 7 days of any active antibiotic treatment from the date of the last positive blood culture
  Interventions: Drug: Short-treatment of any active antibiotic regimen
- Long-treatment of any active antibiotic regimen (Active Comparator): 14 days of any active antibiotic treatment from the date of the last positive blood culture
  Interventions: Drug: Long-treatment of any active antibiotic regimen

INTERVENTIONS:
Drug: Short-treatment of any active antibiotic regimen — 7 days of any active antibiotic treatment for BSI-PA
  Other Names: Any active antibiotic with treatment with proven in vitro activity from a pre-stablished list of antibiotics included
  Arms: Short-treatment of any active antibiotic regimen
Drug: Long-treatment of any active antibiotic regimen — 14 days of any active antibiotic treatment for BSI-PA
  Other Names: Any active antibiotic with treatment with proven in vitro activity a pre-stablished list of antibiotics included
  Arms: Long-treatment of any active antibiotic regimen

SUMMARY:
Phase IV, open-labeled, randomized and multicenter clinical trial to demonstrate the superiority of antibiotics with authorized indication for 7 days versus 14 days in the treatment of bloodstream infections produced by P. aeruginosa (BSI-PA).

DETAILED DESCRIPTION:
The project is designed to determine the optimal duration of antibiotic treatment for Pseudomonas aeruginosa bacteremia, by comparing an adequate antibiotic treatment regimen of 7 days (experimental arm) with another of 14 days (control arm). The evaluation of infection recurrences, mortality, number of free days of antibiotic treatment, adverse events and superinfections are included as secondary objectives.

Active antibiotic treatment will be considered any treatment with proven in vitro activity against the strain responsible for the patient's bacteremia, regardless of the administered dose.

Clinical rules are included in order to stop antibiotic treatment or continuation and re-evaluation in each arm of treatment.

This is a pragmatic study as the number or visits performed for the study are similar to the normal clinical follow-up for this patients. Final contact and final visit for the study will be performed at 90 days after the first positive blood culture.

ELIGIBILITY:
Main inclusion criteria:

* Adult patients with diagnosis of BSI-PA who have received 6 days (+/- 1) of active antibiotic treatment from the date of extraction of the first positive blood culture and until the moment of randomization.
* Informed consent signed.

Main exclusion criteria:

* Bacteremia source not adequately controlled at least 72h before randomization.
* Bacteremia secondary to an infection that necessarily requires prolonged antibiotic treatment more than 7 days
* Coexistence of a different infection at the time of diagnosis of bacteremia that also requires antibiotic treatment.
* Bacteremic pneumonia in severely immunosuppressed patients
* Bacteremia of any origin in patients with severe neutropenia (<500 cells / mm3) at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Probability of achieving better DOOR/RADAR score for patients in the experimental group than in the control group | 30 days after treatment withdrawal
  Probability of any given patient in the experimental arm to achieve better results than a patient in the control group assessed through their score in the DOOR/RADAR ( Desirability of Outcome Ranking/Response Adjusted for Duration of Antibiotic Risk) analysis.
  This analysis categorizes patients in two steps:
  1. A first ordinal clinical outcome ranking (DOOR), defined by the following mutually excluding categories:
     1. Healing without incidences.
     2. Healing with a proven or probable recurrence.
     3. Healing with a serious adverse event.
     4. No clinical cure.
     5. Death.
  2. A second classification in which patients from the same clinical outcome category are ranked according to the number of days of antibiotic treatment (RADAR).
  Patients with a lower DOOR/RADAR score will be those with best outcomes in terms of clinical effectiveness as well as reduced exposure to antibiotic treatment.

SECONDARY OUTCOMES:
Non-inferiority secondary endpoint; Treatment failure | Day +30 from trial treatment interruption
  Defined as mortality from any cause or proven/probable recurrence
Recurrence of infection | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Proven, probable or possible recurrence rate
Mortality from any cause | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Number of patients who died from any cause from the date of inclusion to the final follow-up period
Describe the superinfections | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Superinfection rate
Safety of antibiotic treatment | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture and weighted by 1,000 days of follow-up.
  Gathering any related adverse event from the informed consent form signature up to 90 days
Efficiency of the short-treatment arm | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Number of days of treatment and days of hospital stay avoided at the end of the follow-up period
Confirmation of origin of recurrences | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Checking if the recurrences are due to the same strain, comparing the P. aeruginosa strains by genetic sequencing
Comparison of ecological impact of short and long treatment regimens | Day +30 from trial treatment interruption and day +90 from the date of extraction of the first positive blood culture.
  Diversity of the gut microbiota analysis

CONTACTS AND LOCATIONS:
Overall Officials: José Miguel Cisneros Herreros, MD-PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (37):
- Spain (37):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario de Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario Ciudad de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Final database containing only anonymous data from participant subjects will be shared with direct investigators in a timeframe of 6 months after the complete depuration
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Direct collaborators within the study

REFERENCES:
- [Background] Molina J, Rosso-Fernandez CM, Montero-Mateos E, Pano-Pardo JR, Solla M, Guisado-Gil AB, Alvarez-Marin R, Pachon-Ibanez ME, Gimeno A, Martin-Gutierrez G, Lepe JA, Cisneros JM; SHORTEN-2 trial team. Study protocol for a randomized clinical trial to assess 7 versus 14-days of treatment for Pseudomonas aeruginosa bloodstream infections (SHORTEN-2 trial). PLoS One. 2022 Dec 22;17(12):e0277333. doi: 10.1371/journal.pone.0277333. eCollection 2022. PMID 36548225